CLINICAL TRIAL: NCT04399044
Title: Prophylactic Muscle Flaps for the Prevention of Vascular Graft Infection After Groin Dissection
Brief Title: Prophylactic Muscle Flaps in Vascular Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: per the Institutional Review Board
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2019-1186; A539730 (Other: UW Madison); SMPH/SURGERY/DENTL-PLASTC SRGY (Other: UW Madison); Protocol Version 3/11/2020 (Other: UW Madison)
Record Dates: First submitted 2020-05-18; First posted 2020-05-22 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Vascular Graft Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: No flap (No Intervention): Participants will undergo the scheduled vascular surgery procedure without involvement of the plastic surgery team and use of muscle flaps for graft coverage.
- Group 2: Prophylactic muscle flap (Experimental): Participants will undergo the scheduled vascular surgery procedure and then a muscle flap will be used to cover the vascular graft by a plastic surgeon in the same setting.
  Interventions: Procedure: Prophylactic muscle flap

INTERVENTIONS:
Procedure: Prophylactic muscle flap — A "muscle flap" refers to taking an expendable muscle with its vascular supply and moving it to a new area. In this case, the investigators will take a muscle from the leg or abdomen that is redundant (other muscles perform the same function) and moving it to cover vascular grafts to provide healthy tissue to prevent infection.
  Arms: Group 2: Prophylactic muscle flap

SUMMARY:
Previous studies have suggested that prophylactic muscle coverage in high-risk patients undergoing revascularization procedures through a groin incision have the potential to reduce rates of complications and re-operation. This is a prospective randomized control trial to test this hypothesis at the University of Wisconsin Hospitals and Clinics.

DETAILED DESCRIPTION:
The incidence of graft infections after groin dissection for lower limb revascularization is estimated to be between 2 and 20%. Infection requiring re-operation and muscle flap coverage for salvage is estimated to be between 11 and 13%. Retrospective studies have endeavored to create risk calculators to better predict patients at high risk of need for muscle flap salvage. Fischer et al. suggest that in high-risk patients, prophylactic muscle flaps can reduce complications from 70% to 10%, rates of infection from 70% to 3% and wound breakdown from 48% to 5%. Cost-savings of around $400,000 per year with the use of prophylactic muscle flaps are estimated. Unfortunately, the retrospective nature of the Fischer et al. study, lack of standardization of patients receiving prophylactic muscle flaps, and use of the same cohort for the risk calculator as for the outcomes analysis all reduce the generalizability and reproducibility of these results.

At the University of Wisconsin Hospitals and Clinics, muscle coverage is routinely used in cases of infection or lymph leak but is not systematically used in prophylactic settings. This is because it is generally left to surgeon preference-if they feel like a muscle flap is needed (for a variety of non-standardized anatomic/surgical or patient factors) then it is performed. Muscle coverage of vascular grafts in and of itself is not an experimental procedure and has been performed for decades.

The goal of this study is to determine whether prophylactic muscle flaps in high-risk patients can a) reduce the rates of infection requiring re-operation, and b) reduce the significant morbidity associated with other non-operative complications. This will be the first prospective, randomized control trial to address this issue.

ELIGIBILITY:
Inclusion Criteria:

* Open lower extremity arterial revascularization
* Groin incision
* "High-risk" patients based on risk calculation

Exclusion Criteria:

* Pregnant or breast-feeding
* Any person with diagnosis of an active groin infection preoperatively
* Incarcerated patients
* Unstable patients going directly to the OR for whom the study consent process would delay care, and those who cannot give informed consent to participate in the research study will be excluded
* If a surgeon feels that a patient should or should not receive a flap based on intra-operative or pre-operative characteristics, those patients will be excluded from the study
* Prior to a scheduled groin intervention case a prior authorization will be sent to the participant's insurance company. If the groin flap is denied, which would be highly unusual, then the participant would be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2020-10-16 (Actual); Primary Completion 2021-02-26 (Actual); Study Completion 2021-02-26 (Actual)

PRIMARY OUTCOMES:
Incidence of Graft Infection Requiring Re-operation | within 1 year
  Infection of the vascular graft as determined by clinical diagnosis which requires re-operation for washout or other indicated procedures

SECONDARY OUTCOMES:
Incidence of Infection Not Requiring Re-operation | 1 year
  Superficial infections treated with antibiotics alone or local wound cares
Incidence of Seroma | 1 year
  Fluid collection over the vascular graft
Incidence of Lymphocele | 1 year
  Collection of lymph fluid over vascular graft/operative field
Incidence of Wound Dehiscence | 1year
  Incision breakdown that is managed with wound cares and does not require operative debridement
Toronto Lower Extremity Salvage Score (TESS) at 3 months | 3 months
  This is a 32-item survey of activities commonly performed in daily life, each item scored on a 5 point likert scale where 1 is 'impossible to do' and 5 is 'not at all difficult'. The total possible range of scores is 32 to 160 where higher scores indicate less difficulty in performing tasks. Scores are often standardized to a 100-point scale to account for unanswered questions (referring to activities that they do not normally perform in everyday life).
Toronto Lower Extremity Salvage Score (TESS) at 6 months | 6 months
  This is a 32-item survey of activities commonly performed in daily life, each item scored on a 5 point likert scale where 1 is 'impossible to do' and 5 is 'not at all difficult'. The total possible range of scores is 32 to 160 where higher scores indicate less difficulty in performing tasks. Scores are often standardized to a 100-point scale to account for unanswered questions (referring to activities that they do not normally perform in everyday life).
Toronto Lower Extremity Salvage Score (TESS) at 9 months | 9 months
  This is a 32-item survey of activities commonly performed in daily life, each item scored on a 5 point likert scale where 1 is 'impossible to do' and 5 is 'not at all difficult'. The total possible range of scores is 32 to 160 where higher scores indicate less difficulty in performing tasks. Scores are often standardized to a 100-point scale to account for unanswered questions (referring to activities that they do not normally perform in everyday life).
Toronto Lower Extremity Salvage Score (TESS) at 12 months | 12 months
  This is a 32-item survey of activities commonly performed in daily life, each item scored on a 5 point likert scale where 1 is 'impossible to do' and 5 is 'not at all difficult'. The total possible range of scores is 32 to 160 where higher scores indicate less difficulty in performing tasks. Scores are often standardized to a 100-point scale to account for unanswered questions (referring to activities that they do not normally perform in everyday life).
Readmission rates | 30- and 90-days
  Rates of re-hospitalization after the index revascularization
Total cost of hospitalizations for index diagnosis | 1 year
Number of clinic visits after index surgery | 1 year
Death | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Gast, MD, Study Chair — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Hospital and Clinics, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fischer JP, Nelson JA, Rohrbach JI, Wu LC, Woo EY, Kovach SJ, Low DW, Serletti JM, Kanchwala S. Prophylactic muscle flaps in vascular surgery: the Penn Groin Assessment Scale. Plast Reconstr Surg. 2012 Jun;129(6):940e-949e. doi: 10.1097/PRS.0b013e31824ecb17. PMID 22327893
- [Background] Fischer JP, Nelson JA, Shang EK, Wink JD, Wingate NA, Woo EY, Jackson BM, Kovach SJ, Kanchwala S. Predicting the need for muscle flap salvage after open groin vascular procedures: a clinical assessment tool. J Plast Surg Hand Surg. 2014 Dec;48(6):389-95. doi: 10.3109/2000656X.2014.899242. Epub 2014 Mar 25. PMID 24666001
- [Background] Bennett KM, Levinson H, Scarborough JE, Shortell CK. Validated prediction model for severe groin wound infection after lower extremity revascularization procedures. J Vasc Surg. 2016 Feb;63(2):414-9. doi: 10.1016/j.jvs.2015.08.094. Epub 2015 Oct 30. PMID 26526055